CLINICAL TRIAL: NCT01887574
Title: Renal Mass Registry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-002688
Record Dates: First submitted 2013-06-05; First posted 2013-06-27 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open (Experimental)
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaires given to all patients to assess risk factors and quality of life

SUMMARY:
Collect valuable risk factor and quality of life data from Renal Cell Carcinoma patients and harness the latest technology to organize and analyze data.

DETAILED DESCRIPTION:
RCC is a cancer that is poorly understood. The increase in both incidence and mortality rates for RCC, coupled with the lack of effective therapies for RCC beyond surgical excision, underscore the need for a better understanding of RCC tumor biology, immunology, and epidemiology. Such improved understanding could then be directly translated into new prevention strategies as well as improved patient care. Recently, the National Cancer Institute's Kidney Cancer Progress Review Group identified as top priorities for future research the need to better understand the mechanisms underlying known risk factors for kidney cancer; and examine tumor tissue to identify predictors of patient outcome and targets for therapy. In addition, the review group stressed that the leaders in renal cancer research over the next decade would be those institutions that could enroll large numbers of patients, collect valuable risk factor and quality of life data from these patients and harness the latest technology to organize and analyze data.

ELIGIBILITY:
Inclusion:

* Patients with a renal mass or a suspected metastatic lesion from a renal primary who have been treated or are going to be studied and or treated surgically at Mayo Clinic Arizona
* Patients must be 18 years of age or older
* Patients must be capable of and willing to sign an informed consent

Exclusion:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-06; Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Evidence of Renal Mass Risk Factors as determined by patient questionnaire post surgery | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Erik Castle, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials